CLINICAL TRIAL: NCT01365819
Title: Varenicline for Methamphetamine Dependence: Phase II Clinical Trial
Brief Title: Varenicline for Methamphetamine Dependence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Steve Shoptaw, Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Shoptaw_varen2011
Record Dates: First submitted 2011-05-31; First posted 2011-06-03 (Estimated); Results first posted 2017-02-24 (Actual); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Methamphetamine Dependence; Substance Abuse; Methamphetamine Abuse
Keywords: Crystal meth dependence; crystal meth; methamphetamine dependence; substance abuse
MeSH Terms: conditions — Substance-Related Disorders | interventions — Varenicline; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sugar pill (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Varenicline (Experimental): Varenicline (Chantix (R))
  Interventions: Drug: Varenicline

INTERVENTIONS:
Drug: Varenicline — Varenicline dosing will follow that which has been shown to be effective for cigarette smoking cessation. Varenicline dose will start at 0.5 mg daily for days 1-3, followed by 0.5 mg twice daily for days 4-7, followed by 1 mg twice daily from day 8 until completion of the medication period (end of week 9).
  Other Names: Chantix
  Arms: Varenicline
Drug: Placebo — Placebo dose will start at 0.5 mg (sugar pill) daily for days 1-3, followed by 0.5 mg twice daily for days 4-7, followed by 1 mg twice daily from day 8 until completion of the medication period (end of week 9).
  Other Names: Sugar pill
  Arms: Sugar pill

SUMMARY:
Methamphetamine (MA) dependence is a source of continuing danger for both individuals and society. While there are some behavioral treatments, they are not always effective. To date, there are no medications available to treatment methamphetamine dependence. There is some early evidence suggesting that varenicline (also known as Chantix(tm)) may help people to stop or reduce their use of methamphetamine. Varenicline is already on the market in the U.S. for cigarette smoking cessation and shows promise for treating alcohol dependence. In order to determine if varenicline can help people stop using methamphetamine, we will enroll 90 methamphetamine-dependent people who are looking for treatment into the study at the UCLA Vine Street Clinic operated by Dr Shoptaw of UCLA. Half will receive varenicline (n=45) and half will receive placebo (n=45) which will be determined randomly. Everyone will receive talk therapy for methamphetamine dependence. People will take the medication for 9 weeks followed by a 4 week follow-up period. Before receiving any medication, participants will complete a maximum 2 week (6 study visits) lead-in to complete baseline assessments, psychological and medical evaluation, and comprehensive assessment of drug use to determine study eligibility. If a person is eligible for the study, s/he will receive either varenicline or placebo. Participants will visit the UCLA Vine Street Clinic (UCLA VSC) three times a week study visits. At the end of the medication phase, subjects will complete a four week follow up period for safety monitoring.

DETAILED DESCRIPTION:
Methamphetamine (MA) dependence is a significant source of deleterious consequences to individual and public health including HIV infection, psychological distress, and cardiovascular disease. Behavioral treatments, including cognitive behavioral therapy and contingency management are available, but are modestly effective. Although pharmacotherapy may improve treatment outcomes, ten years of randomized, placebo-controlled trials of medications for MA dependence have failed to identify a medication with a robust effect in generalized populations of MA users.

Cholinergic mechanisms are important in the neurobiology of MA dependence. Varenicline is a α4β2 nicotinic receptor partial agonist and α7 nicotinic receptor full agonist that is approved for cigarette smoking cessation and shows promise for treating alcohol dependence. Varenicline may be effective for the treatment of MA dependence due to: (1) restoration of MA-related dopaminergic deficits via binding to α4β2 receptors in striatal dopaminergic (DA) neurons, (2) reductions in cigarette smoking and the associated nicotine-mediated potentiation of MA effects, (3) activation of the nicotinic cholinergic systems that mediate reductions in reinstatement of MA seeking seen with cannabinoid receptor antagonists and acetylcholinesterase inhibitors, (4) relief of MA-related glutamatergic deficits via α7 nicotinic acetylcholine (ACh) receptor activation, and (5) reduction in MA-related cognitive dysfunction via the cognitive enhancing effects of cholinergic agonists.

The investigators will enroll 90 treatment seeking, MA-dependent participants who will be randomly assigned to receive varenicline (n=45) or placebo (n=45), in conjunction with cognitive behavioral therapy (CBT) for 9 weeks followed by a 4 week follow-up period. Prior to enrollment in the trial, participants will complete a maximum 2 week (6 study visits) lead-in to complete baseline assessments, psychological and medical evaluation, and comprehensive assessment of drug use to determine study eligibility. Once determined to be eligible for the trial, participants will be randomly assigned to varenicline or placebo and will start study medication. Similar to smoking cessation treatment, participants will undergo dose escalation to varenicline 1 mg BID (or placebo BID) over one week as outpatients. Participants will have regular clinic visits at the UCLA Vine Street Clinic (UCLA VSC) for thrice-weekly study visits. At the end of the medication phase, subjects will complete a four-week follow up period for safety monitoring.

ELIGIBILITY:
Inclusion Criteria:

Contact site for additional information.

Exclusion Criteria:

Contact site for additional information.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2012-02; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Shoptaw, PhD, Principal Investigator — UCLA DGSOM Dept Of Family Medicine
Locations (1):
- UCLA Vine Street Clinic, Los Angeles, California, United States

REFERENCES:
- [Background] Zorick T, Sevak RJ, Miotto K, Shoptaw S, Swanson AN, Clement C, De La Garza R 2nd, Newton TF, London ED. Pilot safety evaluation of varenicline for the treatment of methamphetamine dependence. J Exp Pharmacol. 2009 Dec 24;2:13-8. eCollection 2010. PMID 27186086
- [Result] Briones M, Shoptaw S, Cook R, Worley M, Swanson AN, Moody DE, Fang WB, Tsuang J, Furst B, Heinzerling K. Varenicline treatment for methamphetamine dependence: A randomized, double-blind phase II clinical trial. Drug Alcohol Depend. 2018 Aug 1;189:30-36. doi: 10.1016/j.drugalcdep.2018.04.023. Epub 2018 May 25. PMID 29860057

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sugar Pill | Varenicline
Started | 25 | 27
Completed | 12 | 14
Not Completed | 13 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sugar Pill | Varenicline | Total
Number analyzed (Participants) | 25 | 27 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 27 | 52
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 16 | 17 | 33

OUTCOME MEASURES:

1. Primary Outcome: End of Treatment Abstinence
Description: The primary analysis will compare two weeks continuous MA abstinence at end of treatment during weeks 8 and 9 among participants randomly assigned to receive varenicline versus those randomly assigned to receive placebo.
Time Frame: 9 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Sugar Pill | Varenicline
Number analyzed (Participants) | 25 | 27
Participants | 5 | 4

2. Secondary Outcome: Number of Days Retained in Trial
Description: Secondary aims will compare treatment retention among participants randomly assigned to receive varenicline or placebo
Time Frame: 9 weeks
Population: This outcome was not assessed.
Arm/Group | Sugar Pill | Varenicline
Number analyzed (Participants) | 0 | 0

3. Other Pre Specified Outcome: Prevalence of Relapse Following Initiation of Abstinence During Treatment
Description: 1) The number of participants who achieve MA abstinence and subsequently relapse to MA use during treatment by condition (varenicline, placebo) during the outpatient treatment period.
Time Frame: 7 weeks
Population: This analysis presents the number of participants in each condition who achieved abstinence during treatment and later relapsed.
Measure: Count of Participants; unit: Participants
Arm/Group | Sugar Pill | Varenicline
Number analyzed (Participants) | 14 | 13
Participants | 6 | 8

4. Other Pre Specified Outcome: Reduced MA Withdrawal Symptoms
Description: 2) To determine whether varenicline reduces MA withdrawal symptoms more than placebo among MA- dependent participants over the course of the trial.
Time Frame: 9 weeks
Population: This outcome was not assessed.
Arm/Group | Sugar Pill | Varenicline
Number analyzed (Participants) | 0 | 0

5. Other Pre Specified Outcome: Reduction in Cigarette Smoking
Description: 3) To determine whether varenicline reduces cigarette smoking more than placebo among cigarette smoking MA dependent participants.
Time Frame: 9 weeks
Population: This analysis includes a sub-population of participants in both conditions who smoked any cigarettes during treatment. Results are model fitted number of cigarettes smoked per week at baseline and at week 9.
Measure: Mean (Standard Deviation); unit: average number of cigarettes
Units Other Than Participants: average number of cigarettes
Arm/Group | Sugar Pill | Varenicline
Number analyzed (Participants) | 20 | 15
Number analyzed (average number of cigarettes) | 37 | 42
average number of cigarettes | 19 (20) | 1 (3)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the course of the clinical trial, which included 2 weeks of screening, 9 weeks of medication and 4 weeks of follow-up.
Arm/Group | Sugar Pill | Varenicline
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/27
Other Adverse Events (participants affected / at risk) | 17/25 | 21/27
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sugar Pill (N=25) | Varenicline (N=27)
Headache (Nervous system disorders) | 7 (9) | 10 (15)
Insomnia (Psychiatric disorders) | 5 (7) | 9 (11)
Vivid dreams (Psychiatric disorders) | 5 (7) | 12 (15)
Nausea (Gastrointestinal disorders) | 5 (6) | 10 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes